CLINICAL TRIAL: NCT03356561
Title: A Randomized, Double-blind, Placebo-controlled, First-in-Human Phase 1 Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Ad26.ZIKV.001 in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Ad26.ZIKV.001 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108417; VAC26911ZIK1001 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: Ad26.ZIKV.001 5*10^10 Viral Particles (vp) (Experimental): Participants will receive Ad26.ZIKV.001 at 5*10^10 viral particles (vp) via intramuscular (IM) route on Days 1 and 57.
  Interventions: Biological: Ad26.ZIKV.001 5*10^10 vp
- Group 2: Ad26.ZIKV.001 5*10^10 vp and Placebo (Experimental): Participants will receive Ad26.ZIKV.001 5*10^10 vp on Day 1 and placebo on Day 57 via IM route.
  Interventions: Biological: Ad26.ZIKV.001 5*10^10 vp; Biological: Placebo
- Group 3: Ad26.ZIKV.001 1*10^11 vp (Experimental): Participants will receive Ad26.ZIKV.001 at 1*10^11 vp via IM route on Days 1 and 57.
  Interventions: Biological: Ad26.ZIKV.001 1*10^11 vp
- Group 4: Ad26.ZIKV.001 1*10^11 vp and Placebo (Experimental): Participants will receive Ad26.ZIKV.001 1*10^11 vp on Day 1 and placebo on Day 57 via IM route.
  Interventions: Biological: Ad26.ZIKV.001 1*10^11 vp; Biological: Placebo
- Group 5: Placebo (Placebo Comparator): Participants will receive placebo via IM route on Days 1 and 57.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ad26.ZIKV.001 5*10^10 vp — Participants will receive Ad26.ZIKV.001 at a dose of 5*10^10 vp via IM route.
  Other Names: JNJ-66684657
  Arms: Group 1: Ad26.ZIKV.001 5*10^10 Viral Particles (vp); Group 2: Ad26.ZIKV.001 5*10^10 vp and Placebo
Biological: Ad26.ZIKV.001 1*10^11 vp — Participants will receive Ad26.ZIKV.001 at a dose of 1*10^11 vp via IM route.
  Other Names: JNJ-66684657
  Arms: Group 3: Ad26.ZIKV.001 1*10^11 vp; Group 4: Ad26.ZIKV.001 1*10^11 vp and Placebo
Biological: Placebo — Participants will receive placebo via IM route.
  Arms: Group 2: Ad26.ZIKV.001 5*10^10 vp and Placebo; Group 4: Ad26.ZIKV.001 1*10^11 vp and Placebo; Group 5: Placebo

SUMMARY:
The purpose of this study is to assess the safety, reactogenicity, and immunogenicity of Ad26.ZIKV.001 at 2 dose levels, 5*10^10 viral particles (vp) and 1*10^11 vp, administered intramuscularly as single dose and as 2-dose schedules in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy, without significant medical illness, on the basis of physical examination, medical history, and vital signs performed at screening
* Participant must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the laboratory screening tests are outside the laboratory normal reference ranges, and additionally within the limits representing Food and Drug Administration (FDA) toxicity Grade 1, the participant may be considered eligible only if the investigator judges the abnormalities or deviations from normal to be not clinically significant and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participant must agree not to donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after the last study vaccine administration
* Participant must be willing to provide verifiable identification
* All female participants of childbearing potential must have:

  1. a negative serum beta human chorionic gonadotropin (beta-hCG) pregnancy test at screening
  2. a negative urine (beta-hCG) pregnancy test immediately prior to each study vaccine administration

Exclusion Criteria:

* Participant has a known history of flavivirus infection or previous receipt of flavivirus vaccine such as dengue virus (DENV) types 1-4, yellow fever virus (YFV), Japanese encephalitis virus (JEV), and West Nile virus (WNV)
* Participant has traveled to an area with active flavivirus transmission (as per Centers for Disease Control and Prevention [CDC]'s 'Zika travel notices') or Zika cautionary areas ('Yellow and Red areas') within 4 weeks before screening
* Participant has chronic active hepatitis B or hepatitis C virus infection, verified at screening by hepatitis B surface antigen (HBsAg) or hepatitis C antibody, respectively
* Participant has human immunodeficiency virus (HIV) type 1 or type 2 infection
* Participant received or plans to receive licensed live-attenuated vaccines within 28 days before or after each planned study vaccine administration; licensed inactivated, subunit, or conjugate vaccines within 14 days before or after each planned study vaccine administration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-26 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Injection Site (Local) Adverse Events (AEs) | 7 days post vaccination on Day 1 (Day 1 up to Day 8)
  Number of participants with solicited injection site (local) AEs will be evaluated. Solicited local AEs including pain, erythema, and induration at the study vaccine injection site, will be noted in the participant diary from Day 1 to Day 8. Local AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3) and potentially life threatening (Grade 4).
Number of Participants with Solicited Injection Site (Local) Adverse Events (AEs) | 7 days post vaccination on Day 57 (Day 57 up to Day 64)
  Number of participants with solicited injection site (local) AEs will be evaluated. Solicited local AEs including pain, erythema, and induration at the study vaccine injection site, will be noted in the participant diary from Day 57 to Day 64. Local AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3) and potentially life threatening (Grade 4).
Number of Participants with Solicited Systemic AEs | 7 days post vaccination on Day 1 (Day 1 up to Day 8)
  Number of participants with solicited systemic AEs will be evaluated. Following solicited systemic AEs: fever, chills, headache, fatigue, nausea, myalgia, and arthralgia, will be noted in the participant diary from Day 1 to Day 8. Systemic AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3) and potentially life threatening (Grade 4).
Number of Participants with Solicited Systemic AEs | 7 days post vaccination on Day 57 (Day 57 up to Day 64)
  Number of participants with solicited systemic AEs will be evaluated. Following solicited systemic AEs: fever, chills, headache, fatigue, nausea, myalgia, and arthralgia, will be noted in the participant diary from Day 1 to Day 8. Systemic AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3) and potentially life threatening (Grade 4).
Number of Participants with Unsolicited AEs | 28 days post vaccination on Day 1 (Day 1 up to Day 29)
  Number of participants with unsolicited AEs will be evaluated. Unsolicited AEs will include all AEs for which the participant is not specifically questioned in the participant diary. Unsolicited AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3) and potentially life threatening (Grade 4).
Number of Participants with Unsolicited AEs | 28 days post vaccination on Day 57 (Day 57 up to Day 85)
  Number of participants with unsolicited AEs will be evaluated. Unsolicited AEs will include all AEs for which the participant is not specifically questioned in the participant diary. Unsolicited AEs will be graded according to severity as mild (Grade 1), moderate (Grade 2), severe (Grade 3) and potentially life threatening (Grade 4).
Number of Participants with Serious Adverse Events (SAEs) | First vaccination to the end of the study (approximately up to 12 months)
  Number of participants with SAEs will be evaluated. An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant or may require medical or surgical intervention to prevent one of the outcomes listed above.
Number of Participants with Immediate Reportable Events (IREs) | First vaccination to the end of the study (approximately up to 12 months)
  Number of Participants with IREs will be evaluated. Any events of neuroimmunologic significance will be categorized as IREs.

SECONDARY OUTCOMES:
Neutralizing Antibodies to the Vaccine Strain (or Other Strain) | Days 1, 8, 15, 29, 57, 64, 71, 85, 239, and 365
  Zika virus (ZIKV) neutralizing titers of the vaccine-induced immune response will be assessed using a virus neutralization assay (VNA).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (2):
- United States (2):
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Salisch NC, Stephenson KE, Williams K, Cox F, van der Fits L, Heerwegh D, Truyers C, Habets MN, Kanjilal DG, Larocca RA, Abbink P, Liu J, Peter L, Fierro C, De La Barrera RA, Modjarrad K, Zahn RC, Hendriks J, Cahill CP, Leyssen M, Douoguih M, van Hoof J, Schuitemaker H, Barouch DH. A Double-Blind, Randomized, Placebo-Controlled Phase 1 Study of Ad26.ZIKV.001, an Ad26-Vectored Anti-Zika Virus Vaccine. Ann Intern Med. 2021 May;174(5):585-594. doi: 10.7326/M20-5306. Epub 2021 Feb 16. PMID 33587687